CLINICAL TRIAL: NCT00480831
Title: A Randomized, Double-Blind, Phase II Trial of Paclitaxel + Carboplatin + Bevacizumab With or Without PRO95780 in Patients With Previously Untreated, Advanced-Stage Non-Small Cell Lung Cancer
Brief Title: A Study of PRO95780 in Patients With Previously Untreated, Advanced-Stage Non-Small Cell Lung Cancer (APM4074g)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APM4074g
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Cancer; Avastin; APM4074g
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel; drozitumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Drug: PRO95780
- 2 (Placebo Comparator)
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: carboplatin — Intravenous repeating dose
Drug: paclitaxel — Intravenous repeating dose
Drug: placebo — Intravenous repeating dose
  Arms: 2
Drug: PRO95780 — Intravenous repeating dose
  Arms: 1

SUMMARY:
This is a randomized, double-blind, Phase II, placebo-controlled trial adding on to a background of effective treatment designed to evaluate the efficacy, safety, and pharmacokinetics of PRO95780 combined with paclitaxel + carboplatin + bevacizumab therapy in patients with previously untreated Stage IIIB, Stage IV, or recurrent non-small cell lung cancer (NSCLC). Approximately 120 patients will be randomized to one of two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent
* Histologically or cytologically confirmed NSCLC
* Advanced NSCLC
* Measurable disease
* ECOG performance status of 0 or 1
* Age ≥ 18 years
* Use of accepted and effective method of contraception, i.e., double barrier contraceptive methods (e.g., diaphragm plus condom) or abstinence during the course of the study and for 6 months after the last study treatment administration for women, and 1 month for men

Exclusion Criteria:

* Squamous cell histology
* Prior malignancy other than NSCLC (except in situ basal cell carcinoma or in situ cervical cancer), unless it has been treated with curative intent and there is no evidence of disease for ≥ 3 years prior to randomization
* Untreated or unstable CNS metastases
* Myocardial infarction or an unstable or uncontrolled disease or condition related to or impacting cardiac function within 1 year prior to randomization
* Uncontrolled hypertension
* History of arterial thrombosis, stroke, or serious hemorrhagic disorder within 1 year prior to randomization
* Major surgical procedure within 28 days prior to randomization
* Serious non-healing wound ulcer, or bone fracture within 21 days prior to randomization
* Persistent history of gross hemoptysis relating to the patient's NSCLC
* Known HIV infection
* Known to be positive for hepatitis C or hepatitis B surface antigen
* Chronic daily treatment with aspirin or nonsteroidal anti-inflammatory agents known to inhibit platelet function
* Use of anticoagulation therapy
* Participation in clinical trials or undergoing other investigational procedures within 30 days prior to randomization
* Pregnancy (e.g., positive HCG test) or breast feeding
* Known sensitivity to any of the products to be administered during the study
* Any disorder that compromises the ability of the patient to provide written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | Length of study
Changes in vital signs, physical findings, and clinical laboratory results during and following PRO95780 administration | Length of study
Progression-free survival, as determined by independent review facility | Length of study

SECONDARY OUTCOMES:
Objective response and duration of response, as determined by independent review facility | Length of study
Overall survival | 24 months
Progression-free survival, objective response, and duration of objective response, as determined by the investigator | Length of study
Pharmacokinetic parameters | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bray, M.D., Study Director — Genentech, Inc.